CLINICAL TRIAL: NCT03444961
Title: Comprehensive Visual and Mobility Training Using Computer-Assisted Rehabilitation Environment (CAREN) After Argus Retinal Prosthesis Surgery
Brief Title: Computer-Assisted Rehabilitation Environment Training After Argus Retinal Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Aleksandra Rachitskaya, MD, Assistant Professor of Ophthalmology, Cleveland Clinic Lerner College of Medicine, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-1355
Record Dates: First submitted 2017-10-26; First posted 2018-02-26 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Retinitis Pigmentosa
Keywords: Argus II Retinal Prosthesis System; Rehabilitation
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CAREN system training (Experimental): CAREN training
  Interventions: Device: CAREN system training

INTERVENTIONS:
Device: CAREN system training — CAREN allows Argus users to be trained and enhance their device usage in a safe, controlled, and standardized environment.

SUMMARY:
The goal of the current project is to fill the unmet clinical needs around the objective assessment of visual function and develop outcome-oriented visual rehabilitation approach using the computer assisted rehabilitation environment (CAREN) system for Argus recipients.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of the Argus II Retinal Prosthesis System
* Ability to provide informed consent
* Ability to follow two-step commands
* Ability to ambulate 300+ feet with or without visual assistance
* Able to tolerate Argus device turned on for >20 continuous minutes.

Exclusion Criteria:

* Dementia
* Musculoskeletal contraindication to exercise or walking
* Cardiopulmonary contraindication exercise (i.e. uncontrolled heart failure, cardiac arrhythmia, or pulmonary disease).

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Rachitskaya, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rachitskaya A, Yuan A, Davidson S, Streicher M, DeBenedictis M, Rosenfeldt AB, Alberts J. Computer-Assisted Immersive Visual Rehabilitation in Argus II Retinal Prosthesis Recipients. Ophthalmol Retina. 2020 Jun;4(6):613-619. doi: 10.1016/j.oret.2019.11.007. Epub 2019 Nov 15. PMID 31937474

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CAREN System Training
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CAREN System Training
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Effects of CAREN Virtual Reality System on Obstacle Course Navigation
Description: Obstacle course navigation - time (seconds) to complete an obstacle course (walking forward while navigating over a ramp and curb)
Time Frame: 6 wks
Measure: Mean (Full Range); unit: seconds
Groups:
- Pre-CAREN System Training; Post-CAREN Training: CAREN training
  CAREN system training: CAREN allows Argus users to be trained and enhance their device usage in a safe, controlled, and standardized environment.
Arm/Group | Pre-CAREN System Training | Post-CAREN Training
Number analyzed (Participants) | 4 | 4
seconds | 51.25 [28 to 117] | 33.75 [28 to 117]

2. Primary Outcome: Time to Complete the Timed Up and Go Test Before and After CAREN Virtual Reality System Training
Description: Timed Up and Go testing - functional mobility test that requires the individual to stand from a chair, ambulate three meters to a target, turn around, return to the chair, and sit down. Participants were asked to complete two trials was recorded, with a maximum time of 60 seconds per trial.
Time Frame: 6 wks
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Pre - CAREN System Training; Post-CAREN System Training: CAREN training
  CAREN system training: CAREN allows Argus users to be trained and enhance their device usage in a safe, controlled, and standardized environment.
Arm/Group | Pre - CAREN System Training | Post-CAREN System Training
Number analyzed (Participants) | 4 | 4
seconds | 52.8 (6.6) | 39.29 (10.86)

3. Primary Outcome: Effects of CAREN Virtual Reality System on Square Localization Visual Function Test
Description: The square localization test presents a 2.75" square (250 pixels) at a random location on a black background and the patient is instructed to try to touch the square. The test measures the patient's ability to locate an object and results are calculated as a mean error (how far away in pixels from the square the patient touches the screen). A lower mean error (the distance from the square) indicates better patient performance.
Time Frame: 6 wks
Measure: Mean (Full Range); unit: pixels
Arm/Group | Pre-CAREN System Training | Post-CAREN System Training
Number analyzed (Participants) | 4 | 4
pixels | 274.62 [104.12 to 463.47] | 245.43 [104.12 to 463.47]

4. Primary Outcome: Effects of CAREN Virtual Reality System on Direction of Motion Visual Function Test.
Description: The direction of motion test assesses the patient's ability to determine the direction an object is moving. The patient is presented with a white line (1.4'' wide) that moves across the screen in a random series of directions and angles. Patients are instructed to trace their finger on the monitor in the direction they perceived the line moved. Results are calculated as a mean error (how far off, in degrees, was the patient from the direction of the moving line). The higher the mean error/score, the worse the outcome.
Time Frame: 6 wks
Measure: Mean (Full Range); unit: degrees
Arm/Group | Pre-CAREN System Training | Post-CAREN System Training
Number analyzed (Participants) | 4 | 4
degrees | 65.68 [14.51 to 95.16] | 58.12 [14.51 to 95.16]

5. Primary Outcome: Effects of CAREN Virtual Reality System on Grating Visual Acuity Visual Function Test
Description: The grating visual acuity test measures the patient's visual acuity using the principles of acuity charts modified for ultra-low vision subjects. The patients are presented with black and white bars in one of four orientations (horizontal, vertical, diagonal to the left or diagonal to the right). The bars are present on the screen for 5 seconds during which the patient may scan the screen and then provide a verbal response as to which orientation they perceived the bars. The widths of the bars are varied to evaluate different levels of visual acuity. A lower score is associated with better outcomes with 2.9 being the worst possible score.
Time Frame: 6 wks
Measure: Mean (Full Range); unit: logMAR
Arm/Group | CAREN System Training
Number analyzed (Participants) | 4
logMAR | 2.53 [1.7 to 2.9]

6. Primary Outcome: Effects of CAREN Virtual Reality System on Gait Assessment
Description: Subject's gait assessed by meters traveled while localizing objects on the CAREN system. The higher scores are associated with better outcomes (further distance walked).
Time Frame: 6 wks
Measure: Mean (Full Range); unit: meters
Arm/Group | Pre-CAREN System Training | Post-CAREN System Training
Number analyzed (Participants) | 4 | 4
meters | 111.05 [72.84 to 159.70] | 130.7 [72.84 to 159.70]

7. Other Pre Specified Outcome: Effects of CAREN Virtual Reality System on Activities-specific Balance Confidence (ABC) Scale Questionnaire
Description: The Activities-specific Balance Confidence Scale (ABC Scale) is a structured questionnaire that measures an individual's confidence in performing activities without losing balance. It is a 0% to 100% continuous response scale with 0 representing "no confidence" and 100 representing "complete confidence."
Time Frame: 6 wks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Pre-CAREN System Training | Post-CAREN System Training
Number analyzed (Participants) | 4 | 4
units on a scale | 48.125 [0 to 100] | 34.375 [0 to 100]

ADVERSE EVENTS:
Time Frame: AE's were collected over the course of 6 months while patients were enrolled/actively participating in the study.
Arm/Group | CAREN System Training
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03444961/Prot_SAP_000.pdf